CLINICAL TRIAL: NCT02213276
Title: The Effect of Glucose on Bone - Direct or Indirect?
Brief Title: The Effect of Glucose on Bone - Direct og Indirect?
Acronym: GLUBONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-e1
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2014-08

CONDITIONS: Glucose Infusion; Bone Markers; Inflammatory Markers
Keywords: Glucose infusion; Bone markers; Inflammatory markers
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy males (Experimental): Oral glucose tolerance test (OGTT) and intravenous glucose tolerance test (IVGTT).
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: Intravenous Glucose Tolerance Test (IVGTT)

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) — At baseline participants are asked to drink a glucose solution consisting of 75 grams of glucose dissolved in 250 ml of water. Meanwhile and 15 minutes, 30 minutes, 1 hour, 2 hours and 3 hours later, blood is collected from an intravenous access, in order to asses primary and secondary outcomes.
Other: Intravenous Glucose Tolerance Test (IVGTT) — In this intervention, the participant needs to have two intravenous accesses. In one we infuse an adjustable 20% glucose solution, and try to mimic the glucose profile found in the oral glucose tolerance test. In order to do this, blood glucose is measured every 5 minutes. At baseline and 15 minutes, 30 minutes, 1 hour, 2 hours and 3 hours later, blood is collected from another intravenous access, in order to asses primary and secondary outcomes.

SUMMARY:
Diabetes is associated with an increased risk of bone fractures, but current predictors of bone fracture seem to underestimate this risk. It is commonly known that increased levels of certain biochemical bone markers predict low-energy fractures, but the pattern of these markers in diabetics still show heterogeneity and inconsistency. Part of the pathology of diabetes is a high blood glucose level, and this can potentially influence bone turnover and thereby bone markers. Chronic inflammation in patients with inflammatory bowel disease is shown to increase bone resorption, and the same may be the case in diabetics. The purpose of this project is to investigate whether glucose has a direct effect on bone markers or an indirect effect through intestinal hormones or inflammatory processes.

DETAILED DESCRIPTION:
Background

Previous studies have shown that Diabetes Mellitus type I (DMI) and II (DMII) is associated with an increased risk of bone fracture. Paradoxically DMII patients have higher Bone Mineral Density (BMD) than average, while DMI patients have lower BMD than average. Even the low BMD of DMI cannot fully explain the extent of fractures found. Known risk factors and BMD underestimate the risk of fracture amongst DM patients using the 10 year fracture risk tool 'Fracture Risk Assessment Tool' (FRAX). It is well-known that increased levels of biochemical bone markers predict low-energy fractures. However bone markers in DM patients show both heterogeneity and inconsistency. Because of this, the predictive value of bone markers is still uncertain in DM patients. Part of the pathology of DM is a higher blood glucose level than found in non-diabetics. This high level of blood glucose could potentially influence bone turnover and thereby bone markers. It is, however, still uncertain whether glucose per se influences the fracture risk of DM patients. Among young healthy individuals, an Oral Glucose Tolerance Test (OGTT) reduces the concentration of both resorptive and formative bone markers. This reduction can be counteracted by the somatostatin analogue, octreotide. Therefore the effect of glucose on bone markers may be indirect and linked to gut hormone release. It may also be caused by a direct effect on osteocytes or a change in the chemical configuration of bone markers, which render them undetectable by standard assays. To examine this, we have conducted preliminary in vitro trials where glucose was added to serum. This does not change the level of bone markers and it is therefore unthinkable that glucose per se affects the assay or causes changed bone marker configuration. The effect of an Intravenous Glucose Tolerance Test (IVGTT) on bone markers has never been examined. Subcutaneous and parenteral injection of the gut hormone glucagon-like peptide 2 (GLP-2) dose-dependently reduces resorptive bone markers, while parenteral GLP-2 entails no change in formative bone markers. This shows that GLP-2 has an uncoupled effect on bone turnover, where resorption is inhibited, and formation remains the same.

There is an association between bone turnover, inflammation and glucose. Chronic inflammation in patients with inflammatory bowel disease increases bone resorption through an increase in the Receptor Activator of Nuclear factor Kappa beta Ligand/Osteoprotegrin (RANKL/OPG) ratio, and the same may be the case in DMII. Human endothelial cells augment production of the inflammatory marker MCP-1 when glucose levels are continuously elevated. RANKL also induces MCP-1 production in human osteoclasts. An in vitro trial shows, that at blood glucose level of 24 mM, osteoblasts increases expression of RANKL, production of inflammatory markers, including MCP-1, and expression of mRNA for the formative bone marker osteocalcin. It has not yet been examined whether MCP-1 correlates with formative and resorptive bone markers in vivo. It is therefore still uncertain whether glucose has a direct effect on bone turnover or an indirect effect via. either GLP-2 or inflammatory processes.

Aim

The aim of this project is to examine whether IVGTT reduces bone marker levels in the same degree as OGTT does. Also, we examine whether the effect of the glucose load is direct or indirect through either GLP-2 or inflammatory processes reflected by inflammatory markers.

Perspective

This project will determine whether the effect of glucose on bone markers is direct or indirect. This knowledge can then be used to explore whether glucose is 'the missing link' in the present fracture prediction score for DM patients.

Methods

In this project 12 healthy male subjects will undergo both oral glucose tolerance test and intra venous glucose tolerance test. During the tests bone markers will be measured at different time intervals and compared to each other. Using these methods it is possible to distinguish whether glucose acts directly on bone and bone markers or through an intestinal or inflammatory pathway. Subjects will be recruited from advertising. After signing a consent form, subjects will fill out a questionaire concerning lifestyle (smoking, alcohol, diet and exercise), previous fracture and familiar disposition to DM, osteoporosis and thyroid disease. Bloodpressure, height and weight will be measured.

Statistics

Paired t-test and repeated measurement analysis will be used for the statistical analyses, as well as linear and logistical regression for adjustment for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Aged 20 - 50 years

Exclusion Criteria:

* Chronic diseases, including diabetes, but not allergies
* Daily medication use
* Daily dietary supplement use

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The resorptive bone marker S-CTX. | Change from baseline (at 15 minutes, 30 minutes, 1 hour, 2 hours and 3 hours).
  This outcome will be measured for both the oral glucose tolerance test and the intravenous glucose tolerance test, in order to detect differences in bone marker status.
The formative bone marker S-P1NP | Change from baseline (at 15 minutes, 30 minutes, 1 hour, 2 hours and 3 hours).
  This outcome will be measured for both the oral glucose tolerance test and the intravenous glucose tolerance test, in order to detect differences in bone marker status.

SECONDARY OUTCOMES:
S-NTX | Change from baseline (at 15 minutes, 30 minutes, 1 hour, 2 hours and 3 hours).
  Same as for primary outcome.
S-OC | Change from baseline (at 15 minutes, 30 minutes, 1 hour, 2 hours and 3 hours).
  Same as for primary outcome.
RANKL. | Change from baseline (at 15 minutes, 30 minutes, 1 hour, 2 hours and 3 hours).
  Same as for primary outcomes.
Inflammatory markers. | Change from baseline (at 15 minutes, 30 minutes, 1 hour, 2 hours and 3 hours).
  Same as for primary outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Derived] Yan X, Wang Z, Westberg-Rasmussen S, Tarbier M, Rathjen T, Tattikota SG, Peck BCE, Kanke M, Oxvig C, Frystyk J, Starup-Linde J, Sethupathy P, Friedlander MR, Gregersen S, Poy MN. Differential Impact of Glucose Administered Intravenously and Orally on Circulating miR-375 Levels in Human Subjects. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3749-3755. doi: 10.1210/jc.2017-01365. PMID 28973164